CLINICAL TRIAL: NCT00687570
Title: Bowel Preparation With Nutritional Drinks Instead of Traditional Bowel Preparation Before Rectal Cancer Surgery
Brief Title: Bowel Preparation Before Rectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ulf Gustafsson, PhD, MD, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2008/332-31
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Rectal Cancer
Keywords: patients with rectal cancer undergoing surgery; Bowel purity degree; Bowel preparation; Rectal cancer; Nutritional status; complications with traditional bowel preparation; Complications; Physiological status
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Other): Nutritional drinks 7 days before surgery instead of traditional Bowel preparation with Laxabon®
  Interventions: Dietary Supplement: Fresubin Energy Drink
- A (Other): Traditional bowel preparation with Laxabon®
  Interventions: Drug: Laxabon®

INTERVENTIONS:
Dietary Supplement: Fresubin Energy Drink — Fresubin energy drink 30 kcal/kg*dag-1, seven days before surgery
  Arms: B
Drug: Laxabon® — Laxabon® 4 litres starting the day before surgery
  Arms: A

SUMMARY:
Traditionally bowel preparation before surgery of rectal cancer could be troublesome for patients especially for patients with kidney and cardio- vascular diseases, where salt and electrolyte balance can be a problem.

Cleaning the bowel without complications for the patient is one of the aims for this study.

The other aim is to see if patient nutritional status improves with nutritional drinks as a complement to food intake 4-6 weeks before surgery.

DETAILED DESCRIPTION:
In our institution, patients undergoing surgery for cancer in the rectum are often prepared with energy drinks in order to receive a higher energy level before the operation. As a result of this the patients often avoid nausea and have a better intestinal function after surgery and less complications. We think that this treatment has worked well on the patients but no scientific studies have been done on these patients. As a complementary result of the treatment with nutritional drinks we have found that the colon is empty already after a short time of treatment.

The actual study's purpose is to find out if rectal cancer surgery can be performed without traditionally bowel preparation. Nutritional drinks are to be used instead of traditional bowel preparation. Patients are randomized into two groups, stratification for stricture, malnutrition and laparoscopic surgery and each group should either bee treated with traditional bowel preparation, Laxabon® (A) or nutritional drinks, Fresubin Energy drink (B) before surgery. Patients in subgroup B take nutritional drinks seven days before surgery instead of ordinary food. Bowel purity degree is measured peroperatively.

The secondary aim is to see if malnutrition can be improved with nutritional drinks as a complement to ordinary food intake before surgery. For four to six weeks before surgery 50 % or more of the caloric need is substituted with nutritional drinks in subgroup B (Fresubin Energy drink 15-30 kcal/kg*day). Subgroup A only eats ordinary food throughout the same period, before surgery.

Bowel purity degree, physiological functions, and body mass index are measured in all four groups before and after surgery. All patients in the study keep records of physical activity daily, and food diary twice a week. Complications are registered.

Blood samples for hormones and electrolytes are taken before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer
* men
* women
* age 18-90 years

Exclusion Criteria:

* acute ileus
* seriously dementia
* metastatic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Bowel purity degree | day of surgery

SECONDARY OUTCOMES:
Nutritional status | before and after operation
Complications | day of surgery and days after surgery
physiological function | before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Gustafsson, MD, PhD, Principal Investigator — Karolinska Institut
Locations (1):
- Research Department, Ersta Hospital, Stockholm, Sweden